CLINICAL TRIAL: NCT01843660
Title: The Clinical Efficacy and Safety Study of Tramadol Hydrochloride - Paracetamol Tablets in the Treatment of Moderate to Severe Acute Neck-shoulder Pain and Low Back Pain in Orthopaedics Outpatient or Emergency Setting
Brief Title: An Efficacy and Safety Study of Tramadol Hydrochloride-Paracetamol in Treatment of Moderate to Severe Acute Neck-Shoulder Pain and Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016117; TRAMAPPAI4035; TRAMAP-CHN-MA-02
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Results first posted 2013-08-26 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-06

CONDITIONS: Low Back Pain; Shoulder Pain; Neck Pain
Keywords: Low back pain; Shoulder pain; Neck pain; Tramadol hydrochloride; Paracetamol
MeSH Terms: conditions — Low Back Pain; Shoulder Pain; Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tramadol Hydrochloride (HCl)-Paracetamol (Experimental)
  Interventions: Drug: Tramadol HCl-Paracetamol

INTERVENTIONS:
Drug: Tramadol HCl-Paracetamol — Participants will receive 1 to 2 tablets of tramadol HCl-paracetamol orally once daily (each tablet containing tramadol 37.5 milligram [mg] and paracetamol 325mg) for up to a total duration of 6 hours. Additional dose may be given based upon the clinical requirement.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of tramadol hydrochloride-paracetamol tablets in treatment of moderate (medium level of seriousness) to severe (very serious) acute neck, shoulder and low back pain in orthopedics (pertaining to the bones) outpatient or emergency setting.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), non-randomized, multi-center (when more than one hospital or medical school team work on a medical research study) and prospective (study following participants forward in time) study of tramadol hydrochloride-paracetamol tablets. Participants will receive 1 to 2 tablets of tramadol hydrochloride-paracetamol orally once daily (each tablet containing tramadol 37.5 milligram [mg] and paracetamol 325mg). Participants may be given the additional dose according to the clinical requirement. The total treatment duration will be 6 hours. The total study duration will be 4 months. Efficacy will be evaluated primarily by pain intensity and pain relief. Participants will evaluate the pain severity and pain relief at 0.5, 1, 2, 3, 4 and 6 hours respectively after the first dose; and the drug efficacy and overall satisfaction level at the end of 6 hours after the first dose. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Intermittent or persistent pain for less than 3 months, required analgesic therapy, orthopedic surgery and emergency call participants suffering with severe neck, shoulder, low back pain or chronic neck, shoulder, lower back pain, acute (a quick and severe form of illness in its early stage) exacerbation pain
* Pain intensity to be assessed using Numerical Rating Scale (NRS), NRS score more than or equal to 4 (from 0 to 10, 0 = no pain, 10 = extreme pain)
* During normal pain and stable feeling, can study pain assessment methods and can fill in pain control diary
* Be willing to participate in the study and must give written informed consent

Exclusion Criteria:

* Have used strong opium kind of medication 7 days prior to the enrolment
* Have severe mental disease or using antipsychotic (agent that control agitated psychotic behavior, alleviate acute psychotic states, reduce psychotic symptoms, and exert a quieting effect) medication for medical treatment
* Drug abuse/dependence, or chronic alcohol abuse/depend on history
* Pregnant or lactating women
* Unable to tolerate tramadol or any failed treatment in past by using tramadol
* Comparatively more severe pain in other parts of the body than that of the pain mentioned in the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1059 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.

RESULTS

PARTICIPANT FLOW:
Groups:
- Tramadol Hydrochloride (HCl)-Paracetamol: Participants received 1 to 2 tablets of tramadol HCl-paracetamol orally once daily (each tablet containing tramadol 37.5 milligram [mg] and paracetamol 325 mg) for up to a total duration of 6 hours.
Period: Overall Study
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Started | 1059
Completed | 1029
Not Completed | 30
Not completed — Other | 30

BASELINE CHARACTERISTICS:
Population: Out of a total of 1059 participants, baseline characteristic (age and gender) was available for only 1035 participants who were included in the full analysis set.
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Number analyzed (Participants) | 1035
Age Continuous [Mean (Standard Deviation); unit: Years] | 42.43 (12.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 493
  Male | 542

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Score Based on Numeric Rating Scale (NRS) at Hour 0.5
Description: Pain intensity was measured using NRS (0=painless and 10=most severe pain). Score of 1-3 means mild pain; 4-6 means moderate pain and 7-10 means severe pain.
Time Frame: Hour 0.5
Population: Per protocol population included all participants who completed the clinical trial according to the trial protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Number analyzed (Participants) | 1029
Units on a scale | 5.29 (2.07)

2. Primary Outcome: Pain Intensity Score Based on Numeric Rating Scale (NRS) at Hour 1
Description: as for outcome 1
Time Frame: Hour 1
Population: Per protocol population included all participants who completed the clinical trial according to the trial protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Number analyzed (Participants) | 1029
Units on a scale | 4.32 (2.20)

3. Primary Outcome: Pain Intensity Score Based on Numeric Rating Scale (NRS) at Hour 2
Description: as for outcome 1
Time Frame: Hour 2
Population: Per protocol population included all participants who completed the clinical trial according to the trial protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Number analyzed (Participants) | 1029
Units on a scale | 3.52 (2.14)

4. Primary Outcome: Pain Intensity Score Based on Numeric Rating Scale (NRS) at Hour 3
Description: as for outcome 1
Time Frame: Hour 3
Population: Per protocol population included all participants who completed the clinical trial according to the trial protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Number analyzed (Participants) | 1029
Units on a scale | 2.93 (2.00)

5. Primary Outcome: Pain Intensity Score Based on Numeric Rating Scale (NRS) at Hour 4
Description: as for outcome 1
Time Frame: Hour 4
Population: Per protocol population included all participants who completed the clinical trial according to the trial protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Number analyzed (Participants) | 1029
Units on a scale | 2.56 (1.92)

6. Primary Outcome: Pain Intensity Score Based on Numeric Rating Scale (NRS) at Hour 6
Description: as for outcome 1
Time Frame: Hour 6
Population: Per protocol population included all participants who completed the clinical trial according to the trial protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Number analyzed (Participants) | 1029
Units on a scale | 2.39 (1.97)

7. Primary Outcome: Number of Participants With Pain Relief Score at Hour 0.5
Description: Pain relief was measured using 6-point Likert Scale (4=complete, 3=significant/comparatively large, 2=moderate, 1=mild/slight, 0=none, -1=exacerbated/heavier).
Time Frame: Hour 0.5
Population: Per protocol population included all participants who completed the clinical trial according to the trial protocol.
Measure: Number; unit: Participants
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Number analyzed (Participants) | 1029
Participants
  Complete | 7
  Significant | 92
  Moderate | 209
  Mild | 326
  None | 394
  Exacerbated | 1

8. Primary Outcome: Number of Participants With Pain Relief Score at Hour 1
Description: as for outcome 7
Time Frame: Hour 1
Population: Per protocol population included all participants who completed the clinical trial according to the trial protocol.
Measure: Number; unit: Participants
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Number analyzed (Participants) | 1029
Participants
  Complete | 46
  Significant | 226
  Moderate | 271
  Mild | 332
  None | 154
  Exacerbated | 0

9. Primary Outcome: Number of Participants With Pain Relief Score at Hour 2
Description: as for outcome 7
Time Frame: Hour 2
Population: Per protocol population included all participants who completed the clinical trial according to the trial protocol.
Measure: Number; unit: Participants
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Number analyzed (Participants) | 1029
Participants
  Complete | 104
  Significant | 351
  Moderate | 270
  Mild | 230
  None | 74
  Exacerbated | 0

10. Primary Outcome: Number of Participants With Pain Relief Score at Hour 3
Description: as for outcome 7
Time Frame: Hour 3
Population: Per protocol population included all participants who completed the clinical trial according to the trial protocol.
Measure: Number; unit: Participants
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Number analyzed (Participants) | 1029
Participants
  Complete | 179
  Significant | 392
  Moderate | 307
  Mild | 99
  None | 52
  Exacerbated | 0

11. Primary Outcome: Number of Participants With Pain Relief Score at Hour 4
Description: as for outcome 7
Time Frame: Hour 4
Population: Per protocol population included all participants who completed the clinical trial according to the trial protocol.
Measure: Number; unit: Participants
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Number analyzed (Participants) | 1029
Participants
  Complete | 222
  Significant | 484
  Moderate | 194
  Mild | 86
  None | 43
  Exacerbated | 0

12. Primary Outcome: Number of Participants With Pain Relief Score at Hour 6
Description: as for outcome 7
Time Frame: Hour 6
Population: Per protocol population included all participants who completed the clinical trial according to the trial protocol.
Measure: Number; unit: Participants
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Number analyzed (Participants) | 1029
Participants
  Complete | 304
  Significant | 377
  Moderate | 218
  Mild | 78
  None | 51
  Exacerbated | 1

13. Secondary Outcome: Number of Participants Who Required Additional Dosage Administration
Description: Number of participants who additionally required a second tablet within 2 hours after the first administration of the investigational drug was reported.
Time Frame: Baseline up to Hour 2
Population: Per protocol population included all participants who completed the clinical trial according to the trial protocol.
Measure: Number; unit: Participants
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Number analyzed (Participants) | 1029
Participants | 97

14. Secondary Outcome: Number of Participants With Analgesic Satisfaction Score
Description: Participants evaluated their satisfaction with the analgesic effect of the study drug using a 4-point scale (4=very good, 3=good, 2=average, 1=poor). Number of participants in each category was reported.
Time Frame: Hour 6
Population: Per protocol population included all participants who completed the clinical trial according to the trial protocol.
Measure: Number; unit: Participants
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Number analyzed (Participants) | 1029
Participants
  Very good | 128
  Good | 659
  Average | 212
  Poor | 29
  Missing | 1

15. Secondary Outcome: Number of Participants With Overall Analgesic Satisfaction Score
Description: Participants and physicians separately evaluated their satisfaction with the analgesic effect of the study drug using a 5-point scale (1=very unsatisfied, 2 =unsatisfied, 3=average, 4= satisfied and 5=very satisfied). Number of participants in each category was reported.
Time Frame: Hour 6
Population: Per protocol population included all participants who completed the clinical trial according to the trial protocol.
Measure: Number; unit: Participants
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Number analyzed (Participants) | 1029
Participants
  Participants' evaluation: Very unsatisfied | 3
  Participants' evaluation: Unsatisfied | 39
  Participants' evaluation: Average | 207
  Participants' evaluation: Satisfied | 669
  Participants' evaluation: Very satisfied | 111
  Physicians' evaluation: Very unsatisfied | 1
  Physicians' evaluation: Unsatisfied | 33
  Physicians' evaluation: Average | 159
  Physicians' evaluation: Satisfied | 710
  Physicians' evaluation: Very satisfied | 126

ADVERSE EVENTS:
Arm/Group | Tramadol Hydrochloride (HCl)-Paracetamol
Serious Adverse Events (participants affected / at risk) | 0/1059
Other Adverse Events (participants affected / at risk) | 86/1059
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol Hydrochloride (HCl)-Paracetamol (N=1059)
Nausea (General disorders) | 35
Vomiting (General disorders) | 9
Headache (General disorders) | 5
Dizziness (General disorders) | 31
Lethargy (General disorders) | 14
Weakness (General disorders) | 2
Skin itch (General disorders) | 1
Others (General disorders) | 19

LIMITATIONS AND CAVEATS:
Results are reported for 'number of participants who required additional dosage administration' instead of 'time to achieve analgesic effect' due to change in planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction on the PI is that the PI should submit manuscript to the Sponsor for review no less than 60 days prior to public release. Only with written approval of the Sponsor, the results communications could be public released.